CLINICAL TRIAL: NCT05197504
Title: Biomarker Discovery Through Multiomics Study in Advanced Hepatocellular Carcinoma Patients Who Received Atezolizumab and Bevacizumab Combination Therapy
Brief Title: Predictive Biomarkers in Patients With Advanced Hepatocellular Carcinoma Treated With Systemic Therapy
Acronym: HCC
Status: Completed | Type: Observational
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Hong Jae Chon, Assistant professor, Department of Medical Oncology, CHA University
Other Study IDs: 2021-11-019
Record Dates: First submitted 2021-12-24; First posted 2022-01-19 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue, Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- intervention: atezolizumab + bevacizumab
  Interventions: Drug: atezolizumab plus bevacizumab

INTERVENTIONS:
Drug: atezolizumab plus bevacizumab — 1200 mg of atezolizumab plus 15 mg/kg of body weight of bevacizumab intravenously every 3 weeks

SUMMARY:
Hepatocellular carcinoma (HCC) is the third most common cause of cancer-related deaths worldwide, and HCC is more frequently observed in Asia, including South Korea. As HCC is often accompanied by chronic hepatitis B or C virus and liver cirrhosis, treatment of HCC consider not only the tumor but also various factors such as liver function and the patient's performance status. Local treatment and surgery are possible in the early stages of HCC. However, it has a high recurrence rate even after curative surgeries due to underlying cirrhosis and the tumor microenvironment.

Although several studies have investigated gene mutations and differences in treatment response in advanced HCC through next-generation sequencing (NGS), studies on transcriptome analysis of advanced HCC through RNA-sequencing are hard to find, with a need for future research into precise classification and clinical significance of HCC based on multi-omics data.

DETAILED DESCRIPTION:
to establish multi-omics data and discover biomarkers highly associated with treatment response in HCC patients

ELIGIBILITY:
Inclusion Criteria:

* Those above the age of 20 who understand the purpose of the study and agree to participate in the collection of samples during the study.
* Patients who have been diagnosed with unresectable advanced HCC through imaging, histological, or cytological tests.
* Patients who underwent an NGS test with advanced HCC tissues
* Patients who are scheduled to receive systemic treatment
* Patients with measurable lesions based on RECIST v1.1
* ECOG performance status 0 or 1
* Patients with a life expectancy of at least three months

Exclusion Criteria:

* Patients who have systemic conditions accompanied by instability of vital signs, such as infections or organ failure
* Those with mental/neurological conditions or dementia who have difficulties understanding and completing the consent form
* Those who are assessed as not suitable for this study, at the discretion of the researcher

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced HCC will be recruited at CHA Bundang Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
collected tumor samples | through study completion, an average of 3 years
  tumor samples from patients with hepatobiliary cancers (incidence of genetic alteration, association with treatment response and survival duration)
collected blood samples | through study completion, an average of 3 years
  blood samples from patients with hepatobiliary cancers (incidence of genetic alteration, association with treatment response and survival duration)

SECONDARY OUTCOMES:
Multi-omics analysis | 3 years
  Multi-omics analysis to further subtype and find therapeutic targets of HCC
Biomarkers on the efficacy of Atezolizumab+Bevacizumab for advanced HCC | 3 years
  Molecular biomarker associated with overall survival, progression-free survival and objective response rate in patients who receive atezolizumab plus bevacizumab

CONTACTS AND LOCATIONS:
Overall Officials: Hongjae Chon, MD,PhD, Principal Investigator — Principal Investigator
Locations (1):
- CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Background] Zhu AX, Finn RS, Edeline J, Cattan S, Ogasawara S, Palmer D, Verslype C, Zagonel V, Fartoux L, Vogel A, Sarker D, Verset G, Chan SL, Knox J, Daniele B, Webber AL, Ebbinghaus SW, Ma J, Siegel AB, Cheng AL, Kudo M; KEYNOTE-224 investigators. Pembrolizumab in patients with advanced hepatocellular carcinoma previously treated with sorafenib (KEYNOTE-224): a non-randomised, open-label phase 2 trial. Lancet Oncol. 2018 Jul;19(7):940-952. doi: 10.1016/S1470-2045(18)30351-6. Epub 2018 Jun 3. PMID 29875066
- [Background] Finn RS, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Xu DZ, Hernandez S, Liu J, Huang C, Mulla S, Wang Y, Lim HY, Zhu AX, Cheng AL; IMbrave150 Investigators. Atezolizumab plus Bevacizumab in Unresectable Hepatocellular Carcinoma. N Engl J Med. 2020 May 14;382(20):1894-1905. doi: 10.1056/NEJMoa1915745. PMID 32402160
- [Background] Boyault S, Rickman DS, de Reynies A, Balabaud C, Rebouissou S, Jeannot E, Herault A, Saric J, Belghiti J, Franco D, Bioulac-Sage P, Laurent-Puig P, Zucman-Rossi J. Transcriptome classification of HCC is related to gene alterations and to new therapeutic targets. Hepatology. 2007 Jan;45(1):42-52. doi: 10.1002/hep.21467. PMID 17187432
- [Background] Hoshida Y, Toffanin S, Lachenmayer A, Villanueva A, Minguez B, Llovet JM. Molecular classification and novel targets in hepatocellular carcinoma: recent advancements. Semin Liver Dis. 2010 Feb;30(1):35-51. doi: 10.1055/s-0030-1247131. Epub 2010 Feb 19. PMID 20175032
- [Background] Llovet JM, Montal R, Sia D, Finn RS. Molecular therapies and precision medicine for hepatocellular carcinoma. Nat Rev Clin Oncol. 2018 Oct;15(10):599-616. doi: 10.1038/s41571-018-0073-4. PMID 30061739